CLINICAL TRIAL: NCT06125691
Title: A Phase 1, First-in-Human, Randomized, Observer-blind, Controlled, Dose-ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of a Self-Amplifying mRNA Seasonal Influenza Vaccine (ARCT-2138), When Administered to Healthy Adults
Brief Title: Safety and Immunogenicity First-in-human Dose-ranging Study of Self-Amplifying RNA Seasonal Influenza Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Collaborators: Seqirus (Industry); Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARCT-2138-01
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Influenza, Human
Keywords: Influenza; Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Antigens, Surface; Cell Culture Techniques; Aging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Open Label (Part 4 only)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1 of ARCT-2138, younger adults (Experimental): Dose Level 1 of ARCT-2138 administered through intramuscular injection in the deltoid muscle.
  Interventions:
  Investigational Vaccine: ARCT-2138
  Interventions: Biological: ARCT-2138
- Cohort 2 of ARCT-2138, younger adults (Experimental): Dose Level 2 of ARCT-2138 administered through intramuscular injection in the deltoid muscle.
  Interventions:
  Investigational Vaccine: ARCT-2138
  Interventions: Biological: ARCT-2138
- Cohort 3 of ARCT-2138, younger adults (Experimental): Dose Level 3 of ARCT-2138 administered through intramuscular injection in the deltoid muscle.
  Interventions:
  Investigational Vaccine: ARCT-2138
  Interventions: Biological: ARCT-2138
- Cohort 4 of ARCT-2138, younger adults (Experimental): Dose Level 4 of ARCT-2138 administered through intramuscular injection in the deltoid muscle.
  Interventions:
  Investigational Vaccine: ARCT-2138
  Interventions: Biological: ARCT-2138
- Low Dose, younger and older adults (Experimental): Low dose level of ARCT-2138 administered through intramuscular injection in the deltoid muscle.
  Interventions:
  Investigational Vaccine: ARCT-2138
  Interventions: Biological: ARCT-2138
- Medium Dose, younger and older adults (Experimental): Medium dose level of ARCT-2138 administered through intramuscular injection in the deltoid muscle.
  Interventions:
  Investigational Vaccine: ARCT-2138
  Interventions: Biological: ARCT-2138
- High Dose, younger and older adults (Experimental): High dose level of ARCT-2138 administered through intramuscular injection in the deltoid muscle.
  Interventions:
  Investigational Vaccine: ARCT-2138
  Interventions: Biological: ARCT-2138
- Control Dose, younger adults (Active Comparator): Licensed Quadrivalent Vaccine administered through intramuscular injection in the deltoid muscle.
  Interventions:
  Control Vaccine: Licensed Quadrivalent Vaccine for younger adults
  Interventions: Biological: Licensed Quadrivalent Vaccine for younger adults
- Control Dose, older adults (Active Comparator): Licensed Quadrivalent Vaccine administered through intramuscular injection in the deltoid muscle.
  Interventions:
  Control Vaccine: Licensed Quadrivalent Vaccine for older adults
  Interventions: Biological: Licensed Quadrivalent Vaccine for older adults

INTERVENTIONS:
Biological: ARCT-2138 — Each participant will receive one 0.5 mL intramuscular (IM) dose into the deltoid muscle.
  Other Names: Self-Amplifying RNA seasonal Influenza vaccine
  Arms: Cohort 1 of ARCT-2138, younger adults; Cohort 2 of ARCT-2138, younger adults; Cohort 3 of ARCT-2138, younger adults; Cohort 4 of ARCT-2138, younger adults; High Dose, younger and older adults; Low Dose, younger and older adults; Medium Dose, younger and older adults
Biological: Licensed Quadrivalent Vaccine for younger adults — Each participant will receive one 0.5 mL intramuscular (IM) dose into the deltoid muscle.
  Other Names: Influenza vaccine, surface antigen, inactivated, prepared in cell cultures
  Arms: Control Dose, younger adults
Biological: Licensed Quadrivalent Vaccine for older adults — Each participant will receive one 0.5 mL intramuscular (IM) dose into the deltoid muscle.
  Other Names: Influenza vaccine, surface antigen, inactivated, adjuvanted
  Arms: Control Dose, older adults

SUMMARY:
This is a safety and Immunogenicity first-in-human dose-ranging study of self-amplifying RNA Seasonal Influenza Vaccine (ARCT-2138) in adults.

DETAILED DESCRIPTION:
Phase 1, first-in-human, randomized, controlled, observer blind (open label Part 4 only), dose-escalation study, to assess the safety, tolerability, and immunogenicity of different dose levels of the ARCT-2138 vaccine, administered as a single dose to healthy young and older adults, in comparison with an inactivated influenza vaccine.

Study drug (ARCT-2138 or control) will be administered as an intramuscular (IM) injection. The study comprises of four parts. In Part 1, escalating dose levels of ARCT-2138 given as a single injection to younger adults will be evaluated sequentially.

Low, medium, and high dose levels of ARCT-2138 (as recommended by DSMB) will be further evaluated in younger adults in Part 2. Part 3 will evaluate low, medium, and high dose levels of ARCT-2138 (as recommended by DSMB) in older adults.

Part 4 (dose expansion phase) will administer a lower dose of ARCT-2138 in young adults.

Investigational Vaccine: ARCT-2138 (Part 1-3 only, no control vaccine for Part 4) Control Vaccines: licensed influenza vaccines (inactivated)

* For younger adults: Flucelvax® Quad, Seqirus Pty Ltd.
* For older adults: Fluad® Quad, Seqirus Pty Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals are male, female, or transgender adults 18 to 49 years of age or 65 to 85 years of age.
2. Healthy participants or participants with pre-existing stable medical conditions. Pre-existing stable medical condition means a subject who: has full capacity of daily activity and no major medication modification; has not undergone surgical or minimally invasive intervention or had any hospitalization/emergency room visit for the specific medical condition within 3 months prior to Day 1.
3. Participant or legally authorized representatives must freely provide documented informed consent prior to study procedures being performed.
4. Individuals who have not received influenza vaccine within 6 months prior to enrollment.
5. Individuals must agree to comply with all study visits and procedures (including blood tests, nasopharyngeal swabs, diary completion, receipt of telephone calls from the site, willingness to be available for Unscheduled Clinic Visits).
6. Individuals of childbearing potential must be willing to adhere to contraceptive requirements.

Exclusion Criteria:

1. Individuals with acute medical illness or febrile illness, including body temperature >100.4°F (>38.0°C) within 3 days prior to Randomization. These individuals may be offered the opportunity to enter the study after fever and illness has stabilized. Participants with suspected or confirmed influenza should be excluded and referred for medical care. Rescreening will be permitted for individuals who are presented with suspected influenza if another diagnosis is confirmed.
2. Individuals with any medical, neurological, or psychiatric condition that, in the opinion of the investigator, could place the participant at an unacceptable risk of injury or render the participant unable to comply with all study procedures and achieve successful completion of the trial.
3. Individuals with a known history of severe hypersensitivity reactions, including anaphylaxis, or other significant adverse reactions to any mRNA vaccine, influenza vaccine, or excipients.
4. Individuals who have a positive pregnancy test at the Screening visit or Day 1 or who intend to become pregnant or breastfeed during the study.
5. Individuals with a history of myocarditis, pericarditis, myopericarditis or cardiomyopathy.
6. Individuals with a history of Guillain-Barré syndrome, encephalomyelitis, or transverse myelitis.
7. Individuals with a known bleeding disorder that would, in the opinion of the investigator, contraindicate intramuscular (I.M.) injection.
8. Individuals with a history of congenital or acquired immunodeficiency.
9. Individuals who have received immunomodulatory, immunostimulatory, or immunosuppressant drugs including interferon and cytotoxic drugs within 3 months of Screening/Day 1 or who plan to receive them during the study.
10. Individuals requiring systemic corticosteroids exceeding 10 mg/day of prednisone equivalent for ≥10 days within 30 days of Screening. The use of topical, ophthalmic, inhaled, and intranasal steroid preparations will be permitted.
11. Individuals who have received immunoglobulins and/or any blood or blood products within the 3 months before the first vaccine administration or plan to receive such products at any time during the study.
12. Individuals with an immunosuppressive or immunodeficient state, asplenia, or recurrent severe infections.
13. Individuals with a documented history of chronic infection including HIV, HBV, HCV, or who are currently known to have active tuberculosis.
14. Individuals with chronic illness that, in the opinion of the Investigator, are at a stage where it might interfere with trial participation or interpretation of study results.
15. Individuals receiving treatment with another investigational drug, biological agent, or device within 28 days of screening, or 5 half-lives of the investigational drug, whichever is longer; or are currently enrolled in or plan to participate in another clinical trial with an investigational agent during the study period.
16. Individuals who received any influenza vaccine within 6 months prior to enrollment. Individuals who plan to receive an influenza vaccine during the study period*.
17. Individuals who have received any other licensed vaccines within 14 days prior to enrollment in this study or who are planning to receive any vaccine up to 14 days after the study vaccination.
18. Individuals who are investigator site staff members, employees of the Sponsor or the Clinical Research Organization directly involved in the conduct of the study, or site staff members otherwise supervised by the investigator or immediate family members of any of the previously mentioned individuals.

    * Participants in the older adult group (Part 3) are allowed, following their Day 29 visit, to receive the authorized influenza vaccine as per country-specific recommendations.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting local Adverse Events | 14 Days following study vaccination
  Solicited local AEs include injection-site pain, erythema and swelling
Percentage of participants reporting systemic Adverse Events | 14 Days following study vaccination
  Solicited systemic AEs include fatigue, headache, myalgia, arthralgia, nausea, chills, and fever.
Percentage of participants reporting unsolicited Adverse Events | 29 Days following study vaccination
  Spontaneously reported adverse events and as elicited by investigational site staff
Percentage of participants reporting laboratory or vital signs abnormalities | 29 Days following study vaccination
  Abnormal clinically significant values
Percentage of participants reporting serious adverse events, medically attended adverse events adverse events of special interest and adverse events leading early termination | 29 Days following study vaccination
  Spontaneously reported adverse events and as elicited by investigational site staff
Serum hemagglutination inhibition (HAI) antibody levels against the HA glycoprotein. | 29 days following study vaccination
  HAI antibody levels expressed as GMT, GMFI, SCRs and HAI titers.
Serum neuraminidase enzyme-linked lectin (ELLA) assay antibody levels against the NA glycoproteins. | 29 days following study vaccination
  ELLA antibody levels expressed as GMT, GMFI, SCRs and HAI titers.

SECONDARY OUTCOMES:
Percentage of participants reporting serious adverse events, medically attended adverse events adverse events of special interest and adverse events leading early termination | 181 days following study vaccination
  Spontaneously reported adverse events and as elicited by investigational site staff
Serum hemagglutination inhibition (HAI) antibody levels against the HA glycoprotein. | 181 days following study vaccination
  HAI antibody levels expressed as GMT, GMFI, SCRs and HAI titers.
Serum neuraminidase enzyme-linked lectin (ELLA) assay antibody levels against the NA glycoproteins. | 181 days following study vaccination
  ELLA antibody levels expressed as GMT, GMFI, SCRs and HAI titers.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Arcturus Therapeutics
Locations (2):
- Australia (2):
  - Nucleus Network Brisbane Clinic, Brisbane, Queensland
  - Emeritus Research Camberwell, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be made available to study investigators at this time.